CLINICAL TRIAL: NCT07100977
Title: A Randomized, Double-blind, Placebo-controlled, Cross-over Clinical Trial to Investigate the Efficacy of Bragg Apple Cider Vinegar Supplement on Blood Glucose Control in a Healthy Adult Population
Brief Title: A Clinical Trial to Investigate the Acute Effect of Bragg Apple Cider Vinegar Supplement on Blood Glucose Control in a Healthy Adult Population
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bragg Live Food Products (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 25BGCFA02
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-07

CONDITIONS: Postprandial Glucose; Blood Glucose Concentration
Keywords: Apple Cider Vinegar; Apple Cider Vinegar Supplement; Bragg Live Food Products

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bragg ACV Supplement (Experimental): Bragg Apple Cider Vinegar (ACV) Supplement contains apple cider vinegar (standardized to 750 mg of acetic acid), zinc, and vitamin D.
  Interventions: Dietary Supplement: Bragg ACV Supplement
- Placebo (Placebo Comparator): Placebo supplement contains microcrystalline cellulose.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Bragg ACV Supplement — Participants will be instructed to consume 1 capsule of either Bragg ACV Supplement or placebo 10 minutes prior to consumption of a standardized meal.
  Arms: Bragg ACV Supplement
Other: Placebo — Participants will be instructed to consume 1 capsule of either Bragg ACV Supplement or placebo 10 minutes prior to consumption of a standardized meal.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of a Bragg ACV supplement on postprandial glucose excursion compared to a placebo following a standardized acute carbohydrate load.

Participants will be asked to consume an apple cider vinegar supplement 10 minutes prior to a standardized meal.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 20 - 65 years of age, inclusive
2. Females not of child-bearing potential, defined as those who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation) or have been post-menopausal for at least 1 year prior to screening

   Or,

   Individuals of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle and agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner at least 6 months prior to screening
   * Abstinence and agrees to use contraception if planning on becoming sexually active during the study
3. Subjects with elevated fasting glucose > 5.6 mmol/L (> 100 mg/dL) and < 7.0 mmol/L (< 126 mg/dL) and/or elevated HbA1c (6.0-6.4%) and two or more of the other following markers associated with metabolic syndrome at screening:

   1. Abdominal obesity: waist circumference > 102 cm (40 inches) in men and > 88 cm (35 inches) in women
   2. Hypertension: systolic blood pressure > 130 mmHg or diastolic blood pressure > 85 mmHg
   3. Elevated TG: > 150 mg/dL (1.7 mmol/L)
   4. Low HDL-C: < 40 mg/dL (1.03 mmol/L) in men and < 50 mg/dL (1.29 mmol/L) in women
4. Stable body weight defined as a <5% change in body weight in the three months prior to baseline, as assessed by the Qualified Investigator (QI)
5. Agrees to maintain current lifestyle habits (diet, physical activity, medications, supplements, and sleep) as much as possible throughout the study
6. Agrees to comply with dietary guidelines and study requirements prior to in-clinic visits
7. Provided voluntary, written, informed consent to participate in the study
8. Otherwise healthy as determined by medical history and laboratory results as assessed by the Qualified Investigator (QI).

Exclusion Criteria:

1. Individuals who are pregnant, breast feeding, or planning to become pregnant during the study
2. Allergy, sensitivity or intolerance, preventing consumption of investigational product, placebo, or standardized meal
3. Poor venous access as assessed by the QI
4. Current use of prescribed and/or OTC medications, supplements, and/or consumption of food/drinks that may impact the glucose metabolism or efficacy of the investigational product (Sections 7.3.1 and 7.3.2)
5. Unstable metabolic disease or chronic diseases as assessed by the QI
6. Current or history of any significant diseases of the gastrointestinal tract as assessed by the QI
7. Unstable hypertension. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
8. Type I or Type II diabetes
9. Significant cardiovascular event in the past 6 months. Participants with no significant cardiovascular event on stable medication may be included after assessment by the QI on a case-by-case basis
10. History of or current diagnosis with kidney and/or liver diseases as assessed by the QI on a case-by-case basis, with the exception of history of kidney stones in participants who are symptom free for 6 months
11. Self-reported confirmation of current or pre-existing thyroid condition. Treatment on a stable dose of medication for at least 3 months will be considered by the QI
12. Major surgery in the past 3 months or individuals who have planned surgery during the course of the study. Participants with minor surgery will be considered on a case-by-case basis by the QI
13. Cancer, except skin basal cell carcinoma completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable
14. Individuals with an autoimmune disease or are immune compromised as assessed by the QI
15. Self-reported confirmation of a HIV-, Hepatitis B- and/or C-positive diagnosis as assessed by the QI
16. Self-reported confirmation of blood/bleeding disorders as assessed by the QI
17. Chronic inhalation or edible use of cannabinoid products (>1 time/month). Occasional users must agree to abstain from use while participating in the study
18. Regular use of tobacco or nicotine products in the past six months, as assessed by the QI. Occasional users will be required to washout and abstain for the duration of the study period
19. Alcohol intake average of >2 standard drinks per day as assessed by the QI
20. Alcohol or drug abuse within the last 12 months
21. Clinically significant abnormal laboratory results at screening as assessed by the QI
22. Blood donation or blood loss between 101 mL to 449 mL within 30 days prior to screening; blood donation of more than 450 mL within 90 days prior to screening; blood donation during the study or a planned donation within 3 months of the last study visit; or plasma donation (e.g., plasmapheresis) within 15 days prior to screening
23. Participation in other clinical research studies 30 days prior to baseline as assessed by the QI
24. Individuals who are unable to give informed consent
25. Any other condition or lifestyle factor, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
The difference in the incremental area under the curve (iAUC)(0 - 120 min) for venous blood glucose between Bragg ACV supplement and placebo following an acute carbohydrate load. | 0 and 120 minutes post dose
  The difference in the incremental area under the curve (iAUC)(0 - 120 min) for venous blood glucose between Bragg ACV supplement and placebo following an acute carbohydrate load.

SECONDARY OUTCOMES:
The difference between Bragg ACV supplement and placebo following an acute carbohydrate load in the maximum venous blood glucose concentration (Cmax) | 0 and 120 minutes post dose
  The difference between Bragg ACV supplement and placebo following an acute carbohydrate load in the maximum venous blood glucose concentration (Cmax)
The difference between Bragg ACV supplement and placebo following an acute carbohydrate load in the AUC(0 - 120 min) for serum insulin | 0 and 120 minutes post dose
  The difference between Bragg ACV supplement and placebo following an acute carbohydrate load in the AUC(0 - 120 min) for serum insulin
The difference between Bragg ACV supplement and placebo following an acute carbohydrate load in time to maximum concentration for serum insulin (Tmax) | 0 and 120 minutes post dose
  The difference between Bragg ACV supplement and placebo following an acute carbohydrate load in time to maximum concentration for serum insulin (Tmax)

OTHER OUTCOMES:
Incidence of post-emergent adverse events (AE) | Day 0 to 8
  Incidence of post-emergent adverse events (AE)
Clinically relevant changes in blood pressure (BP) after supplementation | Day 0 to 8
  Clinically relevant changes in blood pressure (BP)after supplementation indicating an adverse effect as assessed by the Qualified Investigator
Clinically relevant changes in heart rate (HR) after supplementation | Day 0 to 8
  Clinically relevant changes in heart rate (HR) after supplementation indicating an adverse effect as assessed by the Qualified Investigator

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada